CLINICAL TRIAL: NCT03650985
Title: Diagnosis and Intervention of Complicated Twin Diseases in China
Brief Title: Diagnosis and Intervention of Complicated Twin Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Caixia Liu, Director of the second obstetrical department, Shengjing Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DICTD
Record Dates: First submitted 2018-08-27; First posted 2018-08-29 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Twin Diseases
MeSH Terms: conditions — Diseases in Twins

STUDY DESIGN:
Intervention Model Description: Pregnancy women with complicated twin diseases, who are able to withstand risks of intrauterine treatments and informed consent.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TOCTD (Experimental): Pregnancy women with complicated twin diseases, who are able to withstand risks of intrauterine treatments and informed consent, will be involved. Fetoscope technique will be administered in suitable patients.
  Interventions: Procedure: Fetoscope technique

INTERVENTIONS:
Procedure: Fetoscope technique — Intrauterine intervention with fetoscope technique will be applied to treat complex twin diseases with intention to improve the prognosis of patients.

SUMMARY:
Fetal medicine in China is still a new, young discipline, and the development is very rapid. After nearly 10 years of development, the clinical diagnosis and treatment guidelines of some complicated twin diseases has been established , but they are still needed to be improved. Through this study, the investigators expect to achieve better prediction indicators and early intrauterine precise diagnosis of complicated twin diseases. Also, better procedures of implementing effective intrauterine intervention and assessing the safety and effectiveness of intrauterine intervention are anticipated to be established.

DETAILED DESCRIPTION:
A better guideline for complicated twin diseases are anticipated to be established in China. Molecular genetics and imaging technology are applied to evaluate the outcome and prognosis of intrauterine intervention for complex twin diseases. 3D printing technology is used to assist the preoperative evaluation of fetal intrauterine intervention. Better fetal intrauterine intervention technique and prognosis evaluation are expected to be established.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy women with complicated twin diseases who are able to withstand intrauterine treatment and consent informed.

Exclusion Criteria:

* Pregnancy women who refuse intrauterine treatment.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-08-31 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Gene expression of fetuses | At 20 week of gestational age
  DNA methylation, histone acetylation etc. assessed by analyses of fetal blood and amniotic fluid.
Change of volume of amniotic fluid in Milliliter | At every two week from the sixteenth week of gestational age to delivery of babies
  Measured by doctors of sonography
Change of umbilical artery blood flow | At every two week from the sixteenth week of gestational age to delivery of babies
  Measured by doctors of sonography

SECONDARY OUTCOMES:
Neurodevelopment at early childhood | At age of 1 year old
  Including adaptive, gross motor, fine motor, language, and social function; assessed using Gesell Developmental Schedules.

CONTACTS AND LOCATIONS:
Overall Officials: Caixia Liu, Principal Investigator — Shengjing Hospital
Locations (1):
- Shengjing Hospital, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No